CLINICAL TRIAL: NCT07042880
Title: Facilitating the Assessment of Fundamental Nursing Care in Denmark: Translation, Cultural Adaptation, and Validation of a 41-Item Fundamentals of Care Questionnaire
Brief Title: Cultural Adaptation, and Validation of Fundamentals of Care PRO-tool
Status: Recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: University College Copenhagen (Other)
Responsible Party: Principal Investigator, Maria Kjøller Pedersen, Principal Investigator, Nordsjaellands Hospital
Other Study IDs: NNF24OC0095120
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hospitalized Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
A research team from the University of Seville and Flinders University has created a new 41-item questionnaire to assess fundamental nursing care. This questionnaire focuses on three main areas: the nurse-patient relationship, addressing patients' basic care needs (physical, relational, and psychosocial), and the context of care. This tool helps nurses evaluate and track the quality of care they provide over time.

The questionnaire is a self-administered, patient-reported tool. The questionnaire has been translated into English and adapted for use in Australia, but not yet in Danish. Senior Researcher Maria Kjøller Pedersen from Copenhagen University Hospital, North Zealand is leading the effort to translate and adapt it for Denmark in collaboration with University College Copenhagen.

The goal of this study is to translate, adapt, and validate the questionnaire for use in the Danish healthcare system.

DETAILED DESCRIPTION:
Introduction: A research team from the University of Seville and Flinders University has developed a 41-item questionnaire to assess fundamental nursing care according to the Fundamentals of Care Framework (FoC Intelligence Modelling Tool - FoC-IMT), focusing on the nurse-patient relationship, basic care needs (physical, relational, and psychosocial), and the context of care. This self-administered, patient-reported tool (PRO) helps nurses evaluate and track the patients experience of care over time.

The questionnaire has been translated into English and adapted for use in Australia. Senior Researcher Maria Kjøller Pedersen from Copenhagen University Hospital, North Zealand, is leading the effort to translate and adapt it for Denmark in collaboration with University College Copenhagen. The goal is to translate, adapt, and validate the questionnaire for the Danish healthcare system.

Methods: The study will follow Cruchinho's guideline for translation, cross-cultural adaptation, and validation, comprising eight phases: Forward Translation, Forward Translation Synthesis, Back Translation, Harmonization, Pre-testing, Field Testing, Psychometric Validation, and Psychometric Properties Analysis.

Pre-testing was conducted in a hospital setting. Hospital patients (n=30) and nurses (n=8) were included from Hvidovre Hospital's infection medicine department.

Field testing and validation will be conducted in hospital settings. Hospital patients (n=205) will be recruited from Nordsjællands Hospital's cardiology departments.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for more than 24 hours at a cardiology department

Exclusion Criteria:

* Inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized at cardiology department.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fundamentals of Care | Baseline
  Measured by the Fundamentals of Care Intelligence Modelling Tool

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital, North Zealand, Hillerød
  - Infektionsmedicinsk Afdeling, Hvidovre

IPD SHARING:
Plan to Share IPD: No